CLINICAL TRIAL: NCT01560819
Title: Gut Microbial Transplantation in Pediatric Inflammatory Bowel Diseases
Acronym: GMT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-233
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: ulcerative colitis, gut microbial transplantation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study Participants (Experimental): Participants did not receive any bowel preparation before Gut Microbial Transplantation (GMT). Audio-visual aids were used to help reduce participants' anxiety about GMT.
  Interventions: Drug: Gut Microbial Transplantation

INTERVENTIONS:
Drug: Gut Microbial Transplantation — Each participant received Gut Microbial Transplantation (GMT) as retention enema over a period of 1 hour (60mL enema every 15 minutes) daily for 5 days. Although 240mL of GMT solution was prepared for each participant, the final administered dose was dependent on the subject's comfort and willingness to proceed with the next enema, which was assessed after each enema infusion. Subjects were monitored for 30 minutes after GMT for any immediate adverse events and discharged.
  Other Names: GMT

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic, debilitating, relapsing inflammatory disorder affecting the gastrointestinal tract which does not have a medical cure. IBD consists of 2 different forms: Crohn's Disease (CD) and Ulcerative Colitis (UC). In the last 2 decades, Gut Microbial Transplantation (GMT), also known as fecal transplantation, has been used as a treatment option for Clostridium difficile colitis and UC. The literature supports strong evidence for the plausibility of using GMT for patients with IBD associated colitis, especially for patients with UC.

This research will be conducted in the Helen DeVos Children's Hospital (HDVCH) Pediatric gastrointestinal outpatient clinic. A pilot study of ten patients will be conducted to evaluate if GMT improves clinical symptoms in patients with IBD. Patients with IBD colitis (UC and CD with colonic involvement only) will be approached for GMT as a treatment option for their disease. Each subject will undergo 5 sessions (1 session/day, and not necessarily on consecutive days) of GMT within a period of 10 days. Post treatment evaluation will be done at their regularly scheduled clinic follow up.

Healthy donors >18 years of age will be chosen by the family, inclusive of immediate family members and friends. Donors will be required to complete a screening questionnaire, provide medical history, and undergo blood and stool tests.

ELIGIBILITY:
Participant Inclusion Criteria:

1. Children ages >7 and ≤21 years of age with established diagnosis of Inflammatory Bowel Disease (IBD) colitis (patient with ulcerative colitis (UC) or patients with crohn's disease (CD) with colonic involvement only)
2. Have clinical disease (mild to moderate disease: 10≤ Pediatric Ulcerative Colitis Activity Index (PUCAI) <65)
3. Have stable disease activity and therapy for two months prior to Gut Microbial Transplantation (GMT) procedure.

Participant Exclusion Criteria:

1. Fulminant colitis
2. Indication or scheduled for surgery
3. Pregnancy
4. Use of probiotic supplements during the study period (subjects who have stopped use of probiotic supplements will be eligible as long as they stop taking it 2 weeks prior to Day 1 of GMT)
5. anemia (hemoglobin < 6.0 g/dL) in last one month
6. Graft versus host disease (GVHD)
7. Severely immunocompromised - defined as

   1. History of opportunistic infection (tuberculosis, Pneumocystis jirovecii or systemic fungal infections) in last one year or
   2. Neutropenia: Absolute neutrophil count (ANC) <500
8. Major intra-abdominal surgery within 90 days prior to Day 1 of GMT
9. Administration of any investigational drug within 30 days prior to Day 1 of GMT.
10. Have received infliximab or other tumor necrosis factor (TNF) inhibitors within 2 months prior to Day 1 of GMT or are expected to receive such therapy within 1 month post final GMT.

Donor Inclusion Criteria

1. Based on patient's and parents'/guardian's decision
2. Will be chosen from immediate adult (≥18 years) family members or close friends
3. Should have negative or normal results on screening tests (as explained in donor exclusion criteria below)

Donor Exclusion Criteria (adopted from guidelines provided by American Association of Blood Bank Donor History Questionnaire and American Gastroenterological Association)

1. Positive or abnormal screening test to include:

   1. Hepatitis A Immunoglobulin M (IgM) antibody
   2. Hepatitis B antibody panel suggestive of infection (HBc IgM, HBs Ag, HBs Ab)
   3. Hepatitis C antibody Level
   4. Cytomegalovirus (CMV) IgM antibody
   5. Ebstein Barr Virus (EBV) viral capsid antigen (VCA) IgM antibody
   6. Syphilis Immunoglobulin G (IgG) Ab Screen
   7. Human Immune Deficiency Virus (HIV) I & II enzyme-linked immunosorbent assay (ELISA) screen
   8. Stool i) Fungal smear ii) Stool cultures to exclude Salmonella, Shigella, Escherichia Coli, Campylobacter, Yersinia, Vibrio, Listeria iii) Clostridium difficile toxin assay iv) Ova and parasite screen for Giardia and Cryptosporidium
2. History of metabolic syndrome or gastric bypass surgery
3. History of GI conditions: IBD, irritable bowel syndrome, chronic abdominal pain, GI Malignancy, blood in stool or diarrhea in the last 4 weeks before enrollment
4. Antibiotic or probiotic use within 3 months before enrollment and for the duration of the donation
5. Positive response on screening questionnaire to any of the following:

   1. History of active malignancy or any cancer within the last 5 years (excluding basal cell carcinoma of the skin)
   2. Family history of Creutzfeld-Jacob disease
   3. Corneal or dural transplant
   4. History of high risk sexual behavior (e.g. sexual contact with HIV/acquired immune deficiency syndrome (AIDS) positive, hepatitis positive partner, men who have sex with men, sex for drugs or money)
   5. History of signs of sexually transmitted infections such as genital ulcerations, anogenital herpes, anogenital warts, cancroids or syphilitic lesions
   6. Use of illicit drugs
   7. Travel within the last 6 months to areas of the world where diarrheal illnesses are endemic
   8. History or signs of immunosuppression i) History of any immunosuppressant medication(s) within the last 6 months or history of opportunistic infection(s) in past 1 year ii) Signs of immunosuppression such as:

   <!-- -->

   1. Oral thrush
   2. Disseminated lymphadenopathy

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Kunde, MD, MPH, Principal Investigator — Helen DeVos Children's Hospital of Spectrum Health Hospitals
Locations (1):
- Helen DeVos Children's Hospital of Spectrum Health Hospitals, Grand Rapids, Michigan, United States

REFERENCES:
- [Result] Kunde S, Pham A, Bonczyk S, Crumb T, Duba M, Conrad H Jr, Cloney D, Kugathasan S. Safety, tolerability, and clinical response after fecal transplantation in children and young adults with ulcerative colitis. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):597-601. doi: 10.1097/MPG.0b013e318292fa0d. PMID 23542823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, uncontrolled, single-center, prospective pilot study was conducted at Helen DeVos Children's Hospital's outpatient gastroenterology center. Participants were enrolled between April and December 2012. Each participant took part in the study for 6 weeks. The study was not advertised.
Pre-assignment Details: Fifteen patients with ulcerative colitis (UC) were assessed for eligibility; all showed interest in the study. Ten participants met the eligibility criteria and the donors were identified by the participants.
Groups:
- Study Participants: Ten participants between the ages of 7 to 21 years with mild-to moderate UC (pediatric UC activity index [PUCAI] between 15 and 65) were enrolled in the study. PUCAI is a validated tool to measure disease activity in pediatric UC based on clinical symptoms: a score of <10 = remission; 10-34 = mild disease; 35-64 = moderate disease; 65-85 = severe disease. Participants had stable disease activity and medical treatment for UC for 2 months prior to enrollment. Participants' ongoing treatment for UC was not changed. None of the subjects had concurrent C difficile infection.
- Donors: Healthy donors (>18 years of age) were chosen by the participants. Donors were required to complete a screening questionnaire, provide medical history, and undergo blood and stool tests.
Period: Overall Study
Arm/Group | Study Participants | Donors
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donors: Healthy donors (>18 years of age) were chosen by participants. Donors were required to complete a screening questionnaire, provide medical history, and undergo blood and stool tests.
- Total: Total of all reporting groups
Arm/Group | Study Participants | Donors | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Customized [Mean (Standard Deviation); unit: Years] | 15.2 (4.4) | 39.6 (12.7) | 27.4 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Disease Extent [Number; unit: Participants] — Disease extent: extensive = involving left and transverse colon; left-sided = involving rectum and sigmoid or descending colon; pancolitis = involving the entire colon; proctitis = involving rectum.
  Participants
    Extensive | 1 | 0 | 1
    Left-sided | 1 | 0 | 1
    Pancolitis | 6 | 0 | 6
    Proctitis | 2 | 0 | 2
Disease Activity before Treatment [Number; unit: Participants] — Disease activity: measured by pediatric ulcerative colitis activity index (PUCAI). PUCAI is a validated tool to measure disease activity in pediatric UC based on clinical symptoms: a score of <10 = remission; 10-34 = mild disease; 35-64 = moderate disease; 65-85 = severe disease.
  Participants
    0-9: Remission | 0 | 0 | 0
    10-34: Mild Disease | 3 | 0 | 3
    35-64: Moderate Disease | 7 | 0 | 7
    65-85: Severe Disease | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Clinical response (i.e. improvement in Pediatric Ulcerative Colitis Activity Index (PUCAI) score by greater than or equal to 15 points from baseline) at 4 weeks following GMT treatment
Time Frame: 4 weeks following GMT Treatment
Population: One participant showed intolerance to the treatment (immediate leaking of enema) and was not included in post-treatment disease activity evaluation.
Measure: Number; unit: Participants
Groups:
- Study Participants: Ten participants between the ages of 7 to 21 years with mild-to moderate ulcerative colitis (UC) (pediatric UC activity index [PUCAI] between 15 and 65) were enrolled in the study. PUCAI is a validated tool to measure disease activity in pediatric UC based on clinical symptoms: a score of <10 = remission; 10-34 = mild disease; 35-64 = moderate disease; 65-85 = severe disease. Participants had stable disease activity and medical treatment for UC for 2 months prior to enrollment. Participants' ongoing treatment for UC was not changed. None of the subjects had concurrent C difficile infection.
Arm/Group | Study Participants
Number analyzed (Participants) | 9
Participants | 9
Statistical Analysis 1: Comparison: Study Participants; A power calculation was not done for this pilot study. Changes in PUCAI post-treatment were compared with baseline using the Wilcoxon signed rank test. P value <0.05 was considered statistically significant; Test type: Superiority or Other; p = 0.03, Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded during and until 4 weeks after GMT using a symptom diary that participants completed. Common Terminology Criteria for Adverse Events and Toxicity Grading Guidance from Vaccine Clinical Trials (FDA, 2007) were used.
Description: AEs were collected for study participants, but not donors. Intensity of AEs was classified as mild, moderate, severe, or disabling. AEs were categorized as unrelated or possibly, probably, or definitely related to GMT. Data safety monitoring board was established to monitor AEs and review halting criteria after every 3 participants completed GMT.
Groups:
- Study Participants: Ten participants between the ages of 7 to 21 years with mild-to moderate UC (pediatric UC activity index [PUCAI] between 15 and 65) were enrolled in the study. Participants had stable disease activity and medical treatment for UC for 2 months prior to enrollment. Participants' ongoing treatment for UC was not changed. None of the subjects had concurrent C difficile infection.
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Participants (N=10)
Bloating/flatulance (Gastrointestinal disorders) | 9 (11)
Abdominal pain/cramping (Gastrointestinal disorders) | 6 (11)
Diarrhea (Gastrointestinal disorders) | 6 (9)
Blood in stool (Gastrointestinal disorders) | 3 (5)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This short-term pilot study is limited by its small sample size; therefore, studies with a larger sample size and longer follow-up period will be required to determine true efficacy of GMT in patients with ulcerative colitis (UC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No